CLINICAL TRIAL: NCT06907589
Title: A Novel Accessible and Widespread Healthcare Service Model Based on Technology Innovation for Objective (Early) Diagnosis and Therapeutic Monitoring of Parkinson's Disease Promoting Continuity of Care
Acronym: OLIMPIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scuola Superiore di Studi Universitari e di Perfezionamento Sant'Anna (Other)
Responsible Party: Principal Investigator, Filippo Cavallo, Associate Professor, Scuola Superiore di Studi Universitari e di Perfezionamento Sant'Anna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: OLIMPIA
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease; Healthy Adult
Keywords: parkinson's disease; wearable sensors; motor data
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Data Analysis for Healthy Subjects (Experimental): All subjects who are recruited in the study undergo sensors administration for motor analysis at the enrollement
  Interventions: Device: Motor Data Analysis
- Motor Data Analysis for patients with Parkinson's disease (Experimental): All subjects who are recruited in the study undergo sensors administration for motor analysis at the enrollement
  Interventions: Device: Motor Data Analysis

INTERVENTIONS:
Device: Motor Data Analysis — The SensMode System includes wearable devices for upper and lower limb motion analysis. The upper limb device, SensHand, consists of 3 sensorized elements: 2 sensorized rings to be placed at the level of the distal phalanx of the thumb and forefinger of the hand and 1 sensorized wristband to be placed at the level of the distal portion of the forearm near the wrist. Each element of SensHand allows the acquisition of inertial data with respect to the biomechanics of the arm-forearm-wrist and the first three fingers of the hand, measuring the 3 components in space of linear acceleration, angular velocity, and magnetic field. The lower limb device, SensFoot, is a device that integrates the same electronic components as the bracelet and is placed in a plastic housing shaped like a small rectangular parallelepiped that is placed over the shoe.

SUMMARY:
The present study aims to use the SensMode System - a system composed of wearable devices for upper and lower limb movement analysis and electronic device for data acquisition and processing - on healthy subjects, subjects with idiopathic hyposmia, patients with Parkinson's disease, and subjects with de-novo drug-naïve extrapyramidal syndrome. The purpose is to identify normative data of objective motor measures obtained with such a system, as well as to increase knowledge about the potential contribution such a solution can make to the preclinical diagnosis of Parkinson's disease and the management of patients with this disease.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects - Inclusion Criteria:

   * Adult subjects, both sexes, aged 50-80 years old
   * MMSE score >= 24 absence of olfactory deficit detected on IOIT olfactory test (22). Age class 50-59 years: normal with score <=5; age class 60-69 years: normal with score <=6; age class > 70 years: normal with score <=7
   * absence of neurological diseases
   * absence of functional deficit in the sphere of locomotion as a result of traumatic injury or from other cause to the upper and/or lower limbs and/or pelvis and/or spine
   * expression of informed consent to participate in the study
2. Subjects with Parkinson's disease -- Inclusion criteria:

   * adult subjects, both sexes, 50-80 years of age
   * MMSE score >= 24
   * subjects with Parkinson's disease in the absence of motor fluctuations and dyskinesias, or subjects with Parkinson's disease with mild motor fluctuations throughout the day, but to be examined in the ON phase and in the absence of dyskinesias
   * Hoehn and Yahr stage 1, 2, 3
   * absence of functional deficit in the sphere of locomotion as a result of traumatic injury or from other cause to the upper and/or lower limbs and/or pelvis and/or spine
   * expression of informed consent to participate in the study

Exclusion Criteria:

1. Healthy subjects - Exclusion criteria:

   * denial of informed consent to participate in the study
   * Presence of olfactory deficit detected on IOIT olfactory test. Age class 50-59 years: hyposmia with score >=6; age class 60-69 years: hyposmia with score >=7; age class > 70 years: hyposmia with score >=8
   * body weight greater than 120 kg
   * insufficient degree of cooperation
   * malignant neoplasm in progress or with negative follow-up of less than 6 years
   * structured joint stiffness in the upper and/or lower extremities preventing proper execution of movements
   * paresis and/or plegia of upper and/or lower limb muscle groups from both peripheral and central nerve injury
   * mono/multi/poly sensory and/or motor neuropathy
   * chronic inflammatory diseases with joint involvement of the upper and/or lower limbs
   * vertiginous syndromes in the acute phase
   * neurodegenerative diseases
   * fever
   * venous thrombosis
   * cardiovascular disorders or other acute or chronic conditions capable of affecting the proper performance of motor exercises
   * spinal or joint pain of various etiologies that may affect the performance of motor exercises
   * positive history of recurrent acute cervico-brachialgia and/or lumbosciatica
2. Subjects with Parkinson's disease - Exclusion criteria:

   * Denial of informed consent to participate in the study
   * Hoenn and Yahr stage 4, 5
   * Patient who needs to use an aid (cane or walker) while walking or cannot walk unless aided by a person
   * body weight greater than 120 kg
   * insufficient degree of cooperation
   * malignant neoplasm in place or with negative follow-up of less than 6 years
   * structured joint stiffness in the upper and/or lower extremities that prevents proper execution of movements
   * paresis and/or plegia of upper and/or lower limb muscle groups from both peripheral and central nerve injury mono/multi/poly sensory and/or motor neuropathy
   * chronic inflammatory diseases with joint involvement of the upper and/or lower limbs
   * vertiginous syndromes in the acute phase
   * neurodegenerative diseases, excluding Parkinson's disease
   * fever
   * venous thrombosis
   * cardiovascular disorders or other acute or chronic conditions capable of affecting the proper performance of motor exercises
   * spinal or joint pain of various etiologies that may affect the performance of motor exercises
   * positive history of recurrent acute cervico-brachialgia and/or low back pain

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01-08 (Estimated)

PRIMARY OUTCOMES:
Number of repetitions | at Enrollment (T0)
  Number of repetitions in Finger Tapping task
Number of repetitions | at Enrollment (T0)
  Number of repetitions in Thumb-ForeFinger Tapping task
Number of repetitions | at Enrollment (T0)
  Number of repetitions in Opening/Closing task
Number of repetitions | at Enrollment (T0)
  Number of repetitions in Pronosupination task
Number of repetitions | at Enrollment (T0)
  Number of repetitions in Toe Tapping task
Number of repetitions | at Enrollment (T0)
  Number of repetitions in Leg Agility task
Number of repetitions | at Enrollment (T0)
  Number of repetitions in Heel Tapping task
Number of repetitions | at Enrollment (T0)
  Number of repetitions in Heel-Toe Tapping task
Time to Stand Up | at Enrollment (T0)
  Time to stand up from a chair
Gait Time | at Enrollment (T0)
  Time to walk for 15 meters straight on
Rotation Time | at Enrollment (T0)
  Time to perform a turning of 360°
Fundamental frequency of accelerometer signal | At enrollment (T0)
  Fundamental frequency of accelerometer signal for hands resting tremor task
Fundamental frequency of accelerometer signal | At enrollment (T0)
  Fundamental frequency of accelerometer signal for feet resting tremor task
Fundamental frequency of accelerometer signal | At enrollment (T0)
  Fundamental frequency of accelerometer signal for hands postural tremor task
Fundamental frequency of accelerometer signal | At enrollment (T0)
  Fundamental frequency of accelerometer signal for hands kinetic tremor task
Strides Number | at Enrollment (T0)
  Number of strides to walk for 15 meters straight on

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - Ospedale Santa Maria Annunziata AUSL Toscana Centro, Bagno a Ripoli, Firenze
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - IRCCS Fondazione Don Carlo Gnocchi Firenze, Florence
  - Ospedale Apuane AUSL Toscana Nord Ovest, Massa
  - IRCCS Istituto Auxologico Italiano, Ospedale San Luca, Milan

IPD SHARING:
Plan to Share IPD: No